CLINICAL TRIAL: NCT02731339
Title: Spinal Curvature, Mobility, and Low Back Pain Relationship in Women With and Without Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Seyda TOPRAK CELENAY, Assistant Professor, PT, PhD, Ataturk Training and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2015-31/12
Record Dates: First submitted 2016-03-30; First posted 2016-04-07 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Women with Urinary incontinence (Experimental)
  Interventions: Device: Spinal Mouse® measurement; Behavioral: Low back pain intensity measurement; Behavioral: Urogenital symptoms measurement; Behavioral: Disability caused by low back pain
- Women without Urinary incontinence (Experimental)
  Interventions: Device: Spinal Mouse® measurement; Behavioral: Low back pain intensity measurement; Behavioral: Disability caused by low back pain

INTERVENTIONS:
Device: Spinal Mouse® measurement — The sagittal thoracic spinal curvature and mobility of all participants were assessed with Spinal Mouse® (Idiag, Fehraltorf, Switzerland) in standing position.
Behavioral: Low back pain intensity measurement — Low back pain intensity of the patients was questioned by Visual Analogue Scale
Behavioral: Urogenital symptoms measurement — The presence and severity of various urogenital symptoms was assessed with the Urogenital Distress Inventory-6
  Arms: Women with Urinary incontinence
Behavioral: Disability caused by low back pain — Disability caused by low back pain was assessed with the Oswestry Disability Index

SUMMARY:
The aim of this study was to investigate the relationship among sagittal spinal curvatures, mobility, and low back pain in women with and without urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* aged between 20 and 65 years,
* diagnosed with stress and mixed urinary incontinence
* healthy women

Exclusion Criteria:

* Women with prior history of injury or surgery related to spine,
* spinal deformity,
* systemic pathology,
* any rheumatologic disease,
* neurologic condition,
* symptomatic pelvic organ prolapse,
* malignancy,
* pregnancy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2015-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Spinal curve and mobility, as measured by Spinal Mouse® device | spinal curve and mobility will be followed through study completion, an average of 3 months

SECONDARY OUTCOMES:
Low back pain, as measured by Visual Analog Scale | Low back pain will be followed through study completion, an average of 3 months
Disability caused by low back pain, as measured by Oswestry Disability Index | Disability will be followed through study completion, an average of 3 months
Urogenital symptoms, as measured by Urogenital Distress Inventory-6 | Urogenital symptoms will be followed through study completion, an average of 3 months